CLINICAL TRIAL: NCT01550159
Title: Study of Correlation Between Serum Levels of Markers of Neuronal Injury and Cognitive Dysfunction After Coronary Artery Bypass Graft Surgery
Brief Title: Correlation Between Markers of Neuronal Injury and Cognitive Dysfunction After Coronary Artery Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria José Carvalho Carmona (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Maria José Carvalho Carmona, Study of Correlation Between Serum Levels of Markers of Neuronal Injury and Cognitive Dysfunction after Coronary Artery Bypass Surgery, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 1081/04
Record Dates: First submitted 2012-02-06; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative Cognitive Dysfunction; Cardiac Surgery; General Anesthesia; Neuropsychological Tests
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to evaluate the possible Correlation Between Serum Levels of Markers of Neuronal Injury and Cognitive Dysfunction after Coronary Artery Bypass Surgery.

DETAILED DESCRIPTION:
The systemic inflammatory response after cardiac surgery may cause damage to the central nervous system and elevated markers of brain injury in peripheral blood. This event may be potentially related to the development of postoperative cognitive dysfunction (POCD), with incidences varying from 20 to 83%.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent for coronary artery bypass graft surgery

Exclusion Criteria:

* History of brain disease or dementia, other psychiatric disorders that affect cognition
* Lack of proficiency in Portuguese language

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent for coronary artery bypass graft surgery.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Score in Neuropsycological Tests | 1 year
  Tests for evaluation of quality of life, depressive synths and neuropsycho;logical battery to assess general mental status, learning, attention, visuospatial perception, immediate memory, operational and executive ask and recall, including processing speed. This assessment will be applied before surgery, and 3, 7,21 90 and 180 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maria JC Carmona, MD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- General Hospital of the University od São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva FP, Schmidt AP, Valentin LS, Pinto KO, Zeferino SP, Oses JP, Wiener CD, Otsuki DA, Tort AB, Portela LV, Souza DO, Auler JO Jr, Carmona MJ. S100B protein and neuron-specific enolase as predictors of cognitive dysfunction after coronary artery bypass graft surgery: A prospective observational study. Eur J Anaesthesiol. 2016 Sep;33(9):681-9. doi: 10.1097/EJA.0000000000000450. PMID 27433840